CLINICAL TRIAL: NCT05763823
Title: A Phase 3, Open Label, Single-Arm Clinical Trial to Evaluate the Efficacy and Safety of MK-8228 (Letermovir) for the Prevention of Clinically Significant Cytomegalovirus (CMV) Infection in Chinese Adult, CMV-Seropositive Allogeneic Hematopoietic Stem Cell Transplant Recipients
Brief Title: A Study of Letermovir (MK-8228) to Evaluate Efficacy and Safety for Prevention of Cytomegalovirus Infection in Chinese Hematopoietic Stem Cell Transplant Recipients (MK-8228-045)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8228-045; MK-8228-045 (Other: MSD)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Letermovir (Experimental): Chinese HSCT recipients will receive 240 mg of Letermovir [for participants on Cyclosporin A (CsA)] or 480 mg of Letermovir (for participants not on CsA) either orally or IV once daily through week 14 (~100 days) post-transplant.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Daily 240 mg or 480 mg oral tablets or IV dose
  Other Names: MK-8228

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a once-a-day oral or intravenous (IV) dose of Letermovir (MK-8228) in Chinese adult hematopoietic stem cell transplant (HSCT) recipients for the prevention of clinically significant cytomegalovirus (CMV) infection.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Male/Female Chinese adult participant of an allogeneic Hematopoietic Stem Cell Transplant (HSCT).
* Has documented positive Cytomegalovirus (CMV) serostatus (CMV immunoglobulin G [IgG] seropositive) for recipient (R+) at the time of screening.
* Is receiving a first allogeneic HSCT.
* Is within 28 days post-HSCT at the time of randomization.
* Female participant is not a Woman of Child Bearing Potential (WOCBP) or is a WOBCP who agrees to use acceptable contraception during the treatment period and for ≥28 days after the last dose of study drug.

Exclusion Criteria:

* Received a previous allogeneic HSCT.
* Has a history of CMV end-organ disease within 6 months prior to randomization.
* Has evidence of CMV viremia at any time from HSCT procedure until the time of randomization.
* Has severe hepatic insufficiency.
* Is a) on renal replacement therapy (e.g., hemodialysis, peritoneal dialysis) OR b) has end stage renal impairment with a creatinine clearance <=10 mL/min within 5 days prior to randomization.
* Has both moderate hepatic insufficiency AND moderate to severe renal insufficiency.
* Has an uncontrolled infection on the day of randomization.
* Has rapidly progressing disease that requires mechanical ventilation or is hemodynamically unstable.
* Has a documented positive result for a human immunodeficiency virus antibody (HIV-Ab) test at any time prior to randomization, or for hepatitis C virus antibody (HCV-Ab) with detectable HCV ribonucleic acid (RNA), or hepatitis B surface antigen (HBsAg) within 90 days prior to randomization.
* Has active solid tumor malignancies except localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas).
* Has received any prohibited medications within 2 days prior to initiation of treatment with Letermovir.
* Is anticipated to be treated with Traditional Chinese Medicine or herbal medicine during the study treatment period and for 14 days after study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (21):
- China (21):
  - Anhui Provincial Hospital ( Site 0024), Hefei, Anhui
  - Peking University First Hospital ( Site 0009), Beijing, Beijing Municipality
  - Peking University People's Hospital-Hematology ( Site 0033), Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Third Military Medical University-Oncology Department ( Site 0002), Chongqing, Chongqing Municipality
  - Southwest Hospital of Third Military Medical University ( Site 0005), Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital Chongqing Medical University ( Site 0013), Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital-Hematology Department ( Site 0001), Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital ( Site 0003), Guangzhou, Guangdong
  - Shenzhen Second People's Hospital-Hematology Department ( Site 0006), Shenzhen, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology ( Site 0028), Wuhan, Hubei
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 0032), Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University-hematology department ( Site 0029), Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College ( Site 0022), Xuzhou, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 0021), Nanchang, Jiangxi
  - The First Hospital of Jilin University-Hematology ( Site 0023), Changchun, Jilin
  - The 2nd Affiliated Hospital of Dalian Medical University ( Site 0019), Dalian, Liaoning
  - Shanghai General Hospital ( Site 0018), Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University ( Site 0008), Chengdu, Sichuan
  - The General Hospital of Western Theater Command ( Site 0007), Chengdu, Sichuan
  - Institute of hematology&blood disease hospital-Hematology ( Site 0030), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 0025), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Letermovir: Chinese HSCT recipients received 240 mg of Letermovir [for participants on Cyclosporin A (CsA)] or 480 mg of Letermovir (for participants not on CsA) either orally or IV once daily through week 14 (99 days) post-transplant.
Period: Overall Study
Arm/Group | Letermovir
Started | 120
Completed | 107
Not Completed | 13
Not completed — Death | 6
Not completed — Withdrawal by Parent/Guardian | 1
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Letermovir
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 120
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 120
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Significant Cytomegalovirus (CMV) Infection up to Week 24 Post-Transplant
Description: Clinically significant CMV infection was defined as either one of the following: 1) initiation of anti-CMV pre-emptive therapy based on documented CMV viremia and the clinical condition of the participant or 2) onset of CMV end-organ disease. The percentage of participants with clinically significant CMV infection up to week 24 post-transplant is reported.
Time Frame: Up to Week 24 post-transplant (approximately 6 months)
Population: All allocated participants who received at least 1 dose of study treatment and have no detectable CMV viral deoxyribonucleic acid (DNA) when study intervention is initiated. Per protocol, participants who prematurely discontinued or had a missing outcome at the 24-week visit window were considered treatment failure (i.e. Non-completers equal failure [NC=F] approach was used).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 32 [23.5 to 42.9]

2. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE is reported.
Time Frame: Up to 16 weeks
Population: All allocated participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 120
Percentage of Participants | 99.2 [95.4 to 100.0]

3. Secondary Outcome: Percentage of Participants Who Discontinue Study Treatment Due to an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to 14 weeks
Population: All allocated participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 120
Percentage of Participants | 0 [NA to NA]

4. Secondary Outcome: Percentage of Participants With Clinically Significant CMV Infection up to Week 14 Post-Transplant
Description: Clinically significant CMV infection was defined as either one of the following: 1) initiation of anti-CMV pre-emptive therapy based on documented CMV viremia and the clinical condition of the participant or 2) onset of CMV end-organ disease. The percentage of participants with clinically significant CMV infection up to 14 weeks post-transplant is reported.
Time Frame: Up to 14 weeks post-transplant (99 days)
Population: All allocated participants who received at least 1 dose of study treatment and had no detectable CMV viral DNA when study intervention is initiated. Per protocol, participants who prematurely discontinued or had a missing outcome at the 14-week visit window were considered treatment failure (i.e. Non-completers equal failure [NC=F] approach was used).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 120
Percentage of Participants | 7.1 [2.9 to 14.2]

5. Secondary Outcome: Percentage of Participants With Preemptive Therapy for CMV Viremia up to Week 14 Post-Transplant
Description: Initiation of anti-CMV preemptive therapy was based on documented CMV viremia and the clinical condition of the participant. The percentage of participants with initiation of anti-CMV preemptive anti-CMV therapy up to 14 weeks post-transplant is reported.
Time Frame: Up to 14 weeks post-transplant (99 days)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 7.1 [2.9 to 14.2]

6. Secondary Outcome: Percentage of Participants With Preemptive Therapy for CMV Viremia up to Week 24 Post-Transplant
Description: Initiation of anti-CMV preemptive therapy was based on documented CMV viremia and the clinical condition of the participant. The percentage of participants with initiation of anti-CMV preemptive anti-CMV therapy up to 24 weeks post-transplant is reported.
Time Frame: Up to 24 weeks post-transplant (approximately 6 months)
Population: All allocated participants who received at least 1 dose of study treatment and had no detectable CMV viral DNA when study intervention is initiated. Per protocol, participants who prematurely discontinued or had a missing outcome at the 24-week visit window were considered treatment failure (i.e. Non-completers equal failure [NC=F] approach was used).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 32.7 [23.5 to 42.9]

7. Secondary Outcome: Percentage of Participants With CMV End-organ Disease up to Week 14 Post-Transplant
Description: CMV end-organ disease met per-protocol diagnostic criteria for CMV-pneumonia, gastrointestinal disease, hepatitis, central nervous system disease, retinitis, nephritis, cystitis, myocarditis, pancreatitis, or other disease categories. Only Clinical Adjudication Committee-confirmed CMV end-organ disease will be included in this analysis. The percentage of participants with CMV end-organ disease up to 14 weeks post-transplant is reported.
Time Frame: Up to 14 weeks post-transplant (99 days)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 6.1 [2.3 to 12.9]

8. Secondary Outcome: Percentage of Participants With CMV End-organ Disease up to Week 24 Post-Transplant
Description: CMV end-organ disease met per-protocol diagnostic criteria for CMV-pneumonia, gastrointestinal disease, hepatitis, central nervous system disease, retinitis, nephritis, cystitis, myocarditis, pancreatitis, or other disease categories. Only Clinical Adjudication Committee-confirmed CMV end-organ disease will be included in this analysis. The percentage of participants with CMV end-organ disease up to 24 weeks post-transplant is reported.
Time Frame: Up to 24 weeks post-transplant (approximately 6 months)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 11.2 [5.7 to 19.2]

9. Secondary Outcome: Percentage of Participants With All-Cause Mortality up to Week 14 Post-Transplant
Description: The percentage of participants who died due to any cause up to 14 weeks post-transplant is reported.
Time Frame: Up to 14 weeks post-transplant (99 days)
Population: All allocated participants who received at least 1 dose of study treatment and had no detectable CMV viral DNA when study intervention is initiated.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 5.1 [1.7 to 11.5]

10. Secondary Outcome: Percentage of Participants With All-cause Mortality up to Week 24 Post-Transplant
Description: The percentage of participants who died due to any cause up to 24 weeks post-transplant is reported.
Time Frame: Up to 24 weeks post-transplant (approximately 6 months)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letermovir
Number analyzed (Participants) | 98
Percentage of Participants | 6.1 [2.3 to 12.9]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: All cause mortality is reported for all allocated participants. Serious adverse events and other adverse events are reported for all allocated participants who received at least 1 dose of study treatment.
Arm/Group | Letermovir
All-Cause Mortality (participants affected / at risk) | 8/120
Serious Adverse Events (participants affected / at risk) | 70/120
Other Adverse Events (participants affected / at risk) | 118/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=120)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3)
Dysbiosis (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Sudden cardiac death (General disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3)
Liver injury (Hepatobiliary disorders) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 14 (16)
Acute graft versus host disease in intestine (Immune system disorders) | 4 (4)
Acute graft versus host disease in skin (Immune system disorders) | 1 (2)
Chronic graft versus host disease in intestine (Immune system disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 7 (7)
Cytomegalovirus viraemia (Infections and infestations) | 4 (4)
Epstein-Barr viraemia (Infections and infestations) | 6 (6)
Epstein-Barr virus infection (Infections and infestations) | 8 (8)
Febrile infection (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastrointestinal infection (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 17 (20)
Pneumonia fungal (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute lymphocytic leukaemia refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 12 (12)
Renal failure (Renal and urinary disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=120)
Coagulopathy (Blood and lymphatic system disorders) | 8 (11)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 7 (11)
Abdominal pain upper (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 25 (36)
Haemorrhoids (Gastrointestinal disorders) | 14 (15)
Mouth ulceration (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 27 (32)
Stomatitis (Gastrointestinal disorders) | 11 (13)
Vomiting (Gastrointestinal disorders) | 37 (65)
Asthenia (General disorders) | 8 (9)
Pyrexia (General disorders) | 32 (48)
Hepatic function abnormal (Hepatobiliary disorders) | 13 (14)
Acute graft versus host disease (Immune system disorders) | 16 (16)
COVID-19 (Infections and infestations) | 11 (14)
Conjunctivitis (Infections and infestations) | 9 (9)
Cystitis (Infections and infestations) | 7 (7)
Epstein-Barr virus infection (Infections and infestations) | 20 (27)
Infection (Infections and infestations) | 7 (7)
Pneumonia (Infections and infestations) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 19 (22)
Urinary tract infection (Infections and infestations) | 12 (14)
Alanine aminotransferase increased (Investigations) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 9 (15)
Blood creatinine increased (Investigations) | 8 (13)
Blood lactate dehydrogenase increased (Investigations) | 16 (23)
Gamma-glutamyltransferase increased (Investigations) | 12 (15)
Neutrophil count decreased (Investigations) | 16 (31)
Platelet count decreased (Investigations) | 20 (25)
Weight decreased (Investigations) | 12 (12)
White blood cell count decreased (Investigations) | 27 (53)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9)
Electrolyte imbalance (Metabolism and nutrition disorders) | 10 (11)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (18)
Hyperlipidaemia (Metabolism and nutrition disorders) | 18 (24)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (9)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 16 (23)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 39 (66)
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 20 (36)
Hypoproteinaemia (Metabolism and nutrition disorders) | 19 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 10 (12)
Insomnia (Psychiatric disorders) | 11 (12)
Cystitis haemorrhagic (Renal and urinary disorders) | 19 (19)
Renal failure (Renal and urinary disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 26 (27)
Hypertension (Vascular disorders) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT05763823/Prot_SAP_000.pdf